CLINICAL TRIAL: NCT00538603
Title: Multi-national, Randomized, Phase III, GCIG Intergroup Study Comparing Pegylated Liposomal Doxorubicin (CAELYX) and Carboplatin vs. Paclitaxel and Carboplatin in Patients With Epithelial Ovarian Cancer in Late Relapse. (CALYPSO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC #2051-062
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — liposomal doxorubicin; Carboplatin; CP protocol

INTERVENTIONS:
Drug: pegylated liposomal Doxorubicin (CAELYX) & Carboplatin — Chemotherapy
Drug: Paclitaxel & Carboplatin — Chemotherapy

SUMMARY:
Multi-national, randomized, phase III, GCIG Intergroup study comparing pegylated liposomal Doxorubicin (CAELYX) and Carboplatin vs. Paclitaxel and Carboplatin in patients with epithelial ovarian cancer in late relapse. (CALYPSO)

ELIGIBILITY:
Inclusion Criteria:

* Patients with epithelial Ovarian cancer in late relapse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
overall survival | overall

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Munkarah, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274